CLINICAL TRIAL: NCT02662933
Title: Investigating the Relationship Between Physical Function, Comorbidity and Cytogenetic Risk Group in Older Adults With Acute Myelogenous Leukemia (AML)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00007722; CCCWFU 22A08 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2016-01-19; First posted 2016-01-26 (Estimated); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: ACUTE MYELOGENOUS LEUKEMIA
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bedside Assessment Measures (Experimental): The study intervention consists of a bedside functional assessment to be administered to eligible, consented subjects who are hospitalized with a new diagnosis of AML or are undergoing workup for suspected AML diagnosis. All subjects will be enrolled within 5 days of admission to the hospital for known or suspected AML or within 5 days of new confirmed diagnosis of AML obtained during a hospitalization for other indications. All measures will be performed by a trained examiner during a face to face interview.
  Bedside assessment measures will be repeated once for subjects who complete induction chemotherapy within 2-8 weeks post discharge from initial hospitalization.
  Interventions: Other: Bedside assessment

INTERVENTIONS:
Other: Bedside assessment — The study intervention consists of a bedside functional assessment to be administered to eligible, consented subjects who are hospitalized with a new diagnosis of AML or are undergoing workup for suspected AML diagnosis. All subjects will be enrolled within 5 days of admission to the hospital for known or suspected AML or within 5 days of new confirmed diagnosis of AML obtained during a hospitalization for other indications. All measures will be performed by a trained examiner during a face to face interview.
  Bedside assessment measures will be repeated once for subjects who complete induction chemotherapy within 2-8 weeks post discharge from initial hospitalization.

SUMMARY:
AML is a disease of older adults, with a median age at diagnosis of 67 years . An estimated 13,410 new cases of AML will be diagnosed in 2007. Survival for AML is age-dependent, with significantly lower survival rates reported for older adults. SEER statistics from 1996-2003 show a 5 year relative survival rate of 34.4% for adults younger than 65 and 4.3% for those ≥65 years of age 1. Clinical trials have demonstrated worse survival outcomes in older adults with AML using age cutoffs of 55, 60 and 65 years. Older adults have also experienced increased toxicity to standard therapies in clinical trials. Chronologic age cutoffs have therefore been used in research and clinical practice due to concerns regarding toxicity associated with treatment. The reasons for the increased toxicity and decreased survival in older adults with AML is incompletely understood and likely multifactorial including both tumor specific and host specific factors. Improving understanding of which measurable clinical characteristics predict vulnerability to toxicity will help refine the research and clinical approach to older adults with AML.

ELIGIBILITY:
Inclusion Criteria:

* Capacity to provide signed protocol specific informed consent
* Age ≥ 60 years
* Pathologically confirmed newly diagnosed AML or undergoing workup for suspected AML
* Planned induction chemotherapy
* Inpatient status

Exclusion Criteria:

* Requiring intensive care unit support during initial evaluation
* Prior therapy for AML
* ECOG score >3

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 27 months
  Overall survival will be measured in months from the date of initial AML diagnosis.

SECONDARY OUTCOMES:
Treatment Related Mortality | 30 days
  Treatment-related mortality, defined as death within 30 days of chemotherapy initiation, will provide a general measure of treatment-related toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Klepin, MD, Principal Investigator — Wake Forest University Health Sciences